CLINICAL TRIAL: NCT06648395
Title: Study 2: Testing the Efficacy of a CBT-enhanced Text Message Intervention to Reduce Symptom Burden in Individuals With Post-traumatic Stress Disorder Symptoms and Co-occurring Hazardous Drinking
Brief Title: CBT vs. Supportive Texts for PTSD & Hazardous Drinking (Project Better Study 2)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michele Bedard-Gilligan, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020173; R01AA028776-01A1 (NIH)
Record Dates: First submitted 2024-10-10; First posted 2024-10-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Use; Posttraumatic Stress Disorder
Keywords: Alcohol Use; Posttraumatic Stress Disorder; text messages
MeSH Terms: conditions — Alcohol Drinking; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBT text messages (Active Comparator): Participants in this condition will receive 3 days of text messages for 4 weeks. Day 1 will consist of psychoeducation about a CBT skill, day 2 will be a remainder to use the skill that is framed toward preventing future losses from trauma exposure, and day 3 will have a reminder that aims to instill a growth mindset about using the skill. They will also be asked to complete weekly self-reports on PTSD and HD every Monday for four consecutive weeks.
  Interventions: Behavioral: CBT Text Messages
- Supportive Text Messages (Active Comparator): Participants will be sent three short supportive messages each week that include messages of support, validation, and hope. They will also be asked to complete the weekly self-reports on PTSD and HD every Monday for four consecutive weeks.
  Interventions: Behavioral: Supportive Messages

INTERVENTIONS:
Behavioral: CBT Text Messages — CBT text messages will be sent 3 times per week for 4 weeks
  Arms: CBT text messages
Behavioral: Supportive Messages — Supportive text messages will be sent 3 times per week for 4 weeks
  Arms: Supportive Text Messages

SUMMARY:
The study aims to test the efficacy of a CBT-enhanced text message intervention and a supportive text message intervention to reduce symptom burden in individuals with post-traumatic stress disorder symptoms and co-occurring hazardous drinking.

DETAILED DESCRIPTION:
This study will test a previously piloted and refined text message intervention by comparing a CBT text message intervention to supportive messages condition for reducing hazardous drinking (HD) and PTSD symptoms. The intervention will be tested in a fully powered two-arm randomized controlled trial (RCT) comparing a text message intervention (3 texts/week based on CBT skills) to supportive texts. A sample of 333 participants with DSM-5 Criterion A trauma exposure, PTSD symptoms, and HD will be enrolled and randomized to condition. Baseline, post-, 1-, 3-, 6-, 9-, and 12-month assessments will capture change in primary outcomes (PTSD, hazardous drinking) long-term. Weekly assessments will be given to both conditions to understand shorter-term patterns of symptom change associated with the interventions.

Eligible participants will be individually randomized by the Study Research Coordinator to one of the two conditions. For those in the intervention condition, participants will receive three text messages presenting a CBT skill followed by framing and growth mindsets (sent on Tuesday, Wednesday, Friday). They will also be asked to complete weekly self-reports on PTSD and HD every Monday following their first week of text messages. The supportive messages only group will be sent three short supportive messages, timed to correspond with the CBT skill group, and will be asked to complete the weekly self-reports on PTSD and HD every Monday for four consecutive weeks.

Primary measures include measures assessing inclusion criteria and main outcomes. Primary measures are given at screening/baseline and all follow-ups unless otherwise noted.

Demographics including age, race/ethnicity, gender, income/work status, weight (for BAC calculation for safety monitoring), verification of cell phone ownership and willingness to receive messages, certification of English fluency, and current residential zipcode (to verify WA State residency) will be assessed at screening only.

Trauma exposure and PTSD symptoms will be assessed using the Posttraumatic Stress Disorder Checklist, Civilian Version DSM-5 with the Life Events Checklist (PCL-5 and LEC).

HD will be assessed via a set of measures that provide a detailed picture of drinking patterns. First, two questions will ask about heavy episodic drinking (HED: 4/5 or more drinks per single occasion for men/women) episodes, assessing both frequency over the lifetime and frequency over the last month. Typical weekly alcohol consumption will also be assessed using the Daily Drinking Questionnaire (DDQ). Negative alcohol-related consequences will be assessed via the Short Index of Problems (SIP).

Secondary measures include those assessing secondary outcomes. Unless otherwise noted, secondary measures are given at baseline and 3-, 6-, 9-, and 12-month follow-ups. They include the Alcohol Use Disorders Identification Test (AUDIT), the Depression Anxiety Stress Scales (DASS-21), the Customary Drinking and Drug Use Record (CDDR), the Drug Abuse Screening Test (DAST-10) and the Treatment Services Received (TSR).

Analyses will compare conditions to test effect sizes between the two conditions (text message intervention vs supportive messages). The sample size was selected based on power calculations for detecting a small effect between conditions and also to allow for testing of a-priori chosen effect modifiers (race, gender, trauma type, CBT skill use).

ELIGIBILITY:
Inclusion Criteria:

1. 18+ years of age
2. Currently resides in WA State
3. Fluent in English
4. Reports at least one DSM-5 traumatic event that occurred 1+ months ago
5. Current PTSD severity of 33+ on the PCL-5
6. Current hazardous alcohol use (2+ heavy episodic drinking occasions [4+ drinks on one occasion for women, 5+ drinks on one occasion for men] in past month, 1+ negative consequences related to alcohol use)
7. Owns a functioning cellular phone
8. Is willing to receive weekly study text messages for 4 consecutive weeks
9. Is willing to provide contact information including phone number (for text messages and reminders), email (reminders), and mailing address (payment)

Exclusion Criteria:

1. Previous participation in Project BETTER study 1 (NCT05372042)
2. Participation in Project COPE+ (IRB# STUDY00022875) (a small-scaled text-based message study that aims to increase positive mood and wellbeing for adults with posttraumatic stress symptoms and hazardous drinking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 333 (Estimated)
Dates: Start 2024-10-17 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Posttraumatic Stress Disorder Checklist, Civilian Version DSM-5 (PCL-5) | screening through 12 month follow-up
  The Posttraumatic Stress Disorder Checklist for the 5th Edition of Diagnostic and Statistical Manual of Mental Disorders (PCL-5) assesses the severity of symptoms of posttraumatic stress disorder (PTSD) as defined by the 5th Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and is administered at screening through 12 month follow up. The range of the scale is 0-80. Higher scores represent more severe PTSD symptoms.
Heavy Episodic Drinking (HED) | screening through 12 month follow up
  Heavy Episodic Drinking (HED) assesses the quantity of heavy drinking episodes (i.e., >4/5 drinks per occasion for women/men, based on the National Institute of Alcohol Abuse and Alcoholism's definition) over the last month. It is administered at screening through 12 month follow up. The range of the scale is 0-10 (count of the number of heavy drinking episodes in the last month); 10 is described as 10 or more heavy drinking episodes. Higher scores represent a greater number of heavy drinking episodes.
Daily Drinking Questionnaire (DDQ) | screening through 12 month follow-up
  The Daily Drinking Questionnaire (DDQ) assesses the number of standard drinks consumed each day of a typical week over the last month and is administered at screening through 12 month follow up. The range for the scale to report drinks consumed each day is 0-25. Each day's score for the week is summed to created a total number of drinks consumed per week; the count of drinks consumed per week ranges from 0 to 175. Higher scores representing greater number of drinks consumed during a typical week.
Short Index of Problems (SIP) | screening through 12 month follow-up
  The Short Index of Problems (SIP) assesses the negative consequences from alcohol consumption over the last month and is administered at screening through 12 month follow up. The range for the scale is 0-15. Higher scores represent a greater number of alcohol-related consequences.

SECONDARY OUTCOMES:
Alcohol Use Disorders Identification Test (AUDIT) | screening, 12 month follow-up
  The Alcohol Use Disorders Identification Test (AUDIT) assesses problem drinking and likely diagnosis of an alcohol use disorder over the last 12 months and is administered at pre-intervention (screening) and 12 month follow up. The total range of scores is 0-40. Higher scores represent greater risks of having an alcohol use disorder.
Depression Anxiety Stress Scales (DASS-21) | baseline through 12 month follow-up
  The Depression Anxiety Stress Scale (DASS-21) assesses the general psychopathology symptoms over the last month and is administered at pre-intervention (baseline) through 12 month follow up. It has 3 subscales; two of which (anxiety and depression subscales) are outcomes for this study. The total range of scores of the anxiety subscale of the DASS-21 is 0-21 and higher scores indicate more severe symptoms. The total range of scores of the depression subscale of the DASS-21 is 0-21 and higher scores indicate more severe symptoms.
Customary Drinking and Drug Use Record (CDDR) | baseline, 12 month follow-up
  The Customary Drinking and Drug Use Record (CDDR) assesses comprehensive substance use, other than alcohol, over the last 3 months and is administered at pre-intervention (baseline) and 12 month follow up. The total range of scores is 0-12 and higher scores indicate more drug use.
Drug Abuse Screening Test (DAST-10) | baseline, 12 month follow-up
  The Drug Abuse Screening Test (DAST-10) assesses the problems related to other substance use and likely drug use disorder diagnosis over the last 12 months and is administered at pre-intervention (baseline) and 12 month follow up. The total range of scores is 0-10 and higher scores indicate more substance use-related problems and likely drug use disorder diagnosis.
Treatment Services Received (TSR) | baseline and 12 month follow-up
  The Treatment Services Received (TSR) assesses the types of mental health and addictions treatments that individuals (e.g., inpatient, outpatient, 12-step, etc) received since enrolling in the study and is administered at pre-intervention (baseline) and 12 month follow up. Twelve types of treatment are listed and counted to calculate the number of types of treatment that individuals received over the study period. The minimum possible score is 0 (no services received) and the maximum is 12 types of treatment. Higher numbers indicate receiving more types of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Lindgren, PhD, ABPP, Principal Investigator — University of Washington; Michele Bedard-Gilligan, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bedard-Gilligan M, Lindgren K, Dworkin E, Tristao T, Kaysen D, Rhew I. A randomized controlled trial testing theory-driven enhancements to increase the efficacy of and engagement in a brief cognitive-behavioural therapy text-message intervention for co-occurring posttraumatic stress disorder symptoms and alcohol misuse. Br J Clin Psychol. 2025 Mar;64(1):110-124. doi: 10.1111/bjc.12463. Epub 2024 Mar 26. PMID 38532251
- [Background] Bedard-Gilligan MA, Dworkin ER, Kaysen D, Ojalehto HJ, Stappenbeck CA, Lindgren KP. A pilot study on the feasibility, acceptability, and preliminary efficacy of a brief text message intervention for co-occurring alcohol misuse and PTSD symptoms in a community sample. J Anxiety Disord. 2022 Oct;91:102615. doi: 10.1016/j.janxdis.2022.102615. Epub 2022 Aug 6. PMID 35988440